CLINICAL TRIAL: NCT04910854
Title: A Study of Surufatinib in the Treatment of Recurrent/Metastatic Adenocarcinomas of the Head and Neck
Brief Title: Surufatinib in Recurrent/Metastatic Head and Neck Adenocarcinomas
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021HNRT02
Record Dates: First submitted 2021-05-28; First posted 2021-06-02 (Actual); Last update posted 2021-06-02 (Actual); Status verified 2021-05

CONDITIONS: Head and Neck Cancers - Salivary Gland
MeSH Terms: interventions — surufatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Surufatinib — Patients receive oral Surufatinib at a dose of 300mg/d (once-daily dosing continuously, every 28-day treatment cycle), The curative effect was evaluated every 8 weeks.

SUMMARY:
This is a non-randomized, phase II, open label study of Surufatinib hydrochloride capsules in recurrent/metastatic adenocarcinomas of head and neck. The primary purpose of this study is to evaluate the efficacy of anlotinib.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of written Informed Consent Form (ICF) prior to any study specific procedures;
2. Male and Female aged between 18 and 75 years are eligible;
3. Histologically or cytologically confirmed that recurrent or metastatic adenocarcinomas of the head and neck;
4. Patients with recurrent or metastatic head and neck adenocarcinoma who are not candidates for curative surgery or refusing surgical treatment;
5. Presence of at least one measurable target lesion for further evaluation according to RECIST criteria;
6. Eastern Cooperative Oncology Group (ECOG) performance status 0-2;
7. Predicted survival ≥6 months;
8. Screening laboratory values must meet the following criteria (within past 14 days):

   * neutrophils ≥1.5×109/L ;
   * platelets ≥9g/dL；
   * hemoglobin ≥ 9.0 g/dL;
   * albumin≥3g/dL；
   * total bilirubin ≤ 1.5 x upper limit of normal (ULN); aspartic transaminase (AST) and alanine transaminase (ALT) ≤ 2.5 x ULN without, and ≤ 5 x ULN with hepatic metastasis; serum creatinine ≤1.5╳ULN;
9. Males or female of childbearing potential must: agree to use using a reliable form of contraception (eg, oral contraceptives, intrauterine device, control sex desire, double barrier method of condom and spermicidal) during the treatment period and for at least 6 months after the last dose of study drug.

Exclusion Criteria:

* 1. Prior treatment with Surufatinib,or other antiangiogenic drugs were used within 6 months; 2. Prior antitumor therapy with chemotherapy, radical radiation therapy ，biological immunotherapy，targeted therapy within 4 weeks.

  3. Prior participation in other clinical trials not approved or listed in China within past 4 weeks； 4. Prior major surgery within past 4 weeks (diagnostic surgery excluded); 5. International standardized ratio (INR) >1.5 or partially activated prothrombin time (APTT) >1.5×ULN; 6. Clinically significant severe electrolyte abnormality judged by investigator ; 7. Hypertension that is not controlled by the drug, and is defined as: SBP≥140 mmHg and/or DBP≥90 mmHg; 8. Currently suffering from poorly controlled diabetes (after regular treatment, fasting plasma glucose concentration ≥10mmol/L); 9. The patient currently has disease or condition that affects the absorption of the drug, or the patient cannot be administered orally; 10. Digestive tract disease such as gastric and duodenal active ulcer, ulcerative colitis or unresected tumor, or other conditions determined by the investigator that may cause gastrointestinal bleeding and perforation; 11. Evidence of bleeding tendency or history within 3 months, or thromboembolic event (including a stroke event and/or a transient ischemic attack) occurred within 12 month; 12. Cardiovascular disease of significant clinical significance (myocardial infarction, unstable arrhythmia or unstable angina ，Coronary Artery Bypass Grafting within past 6 months,)； 13. Had other malignant tumors in the past 5 years (except for basal cell carcinoma or squamous cell carcinoma, cervical carcinoma in situ that have been effectively controlled); 14. Active or uncontrolled severe infection (≥CTCAE2 infection); 15. Positive tests for HIV, HCV, HBsAg or HBcAb with positive test for HBV DNA (>2000IU/ml); 16. Evidence with active CNS disease or previous brain metastases; 17. The toxicity associated with previous anti-tumor treatment has not recovered to ≤CTCAE1, except for peripheral neurotoxicity and alopecia ≤CTCAE2 caused by oxaliplatin; 18. Pregnant or nursing; 19. Transfusion therapy, blood products and hematopoietic factors, such as albumin and granulocyte colony stimulating factor (G-CSF), had been received within 14 days before enrollment; 20. Tumor involving skin and/or pharyngeal mucosa with ulceration; 21. Patients with a history of psychotropic drug abuse and unable to quit or with mental disorders; 22. Any other disease, with clinical significance of metabolic abnormalities, abnormal physical examination or laboratory abnormalities, according to researchers, there is reason to doubt is not suitable for the use of study drugs in patients with a disease or condition (such as have a seizure and require treatment), or will affect the interpretation of results, or make the patients at high risk.

  23. Routine urine indicated that urine protein ≥2+, and the 24-hour urine protein volume >1.0g; 24. Underlying medical condition that, in the Investigator's opinion, would increase the risks of study drug administration or obscure the interpretation of toxicity determination or adverse events.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-03-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | up to 24 months

SECONDARY OUTCOMES:
Disease Control Rate (DCR） | up to 24 months
Progress free survival (PFS) | up to 24 months
Overall Survival (OS) | up to 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No